CLINICAL TRIAL: NCT00569270
Title: Simplified Detection of Dynamic Hyperinflation Using Metronome Paced Hyperventilation and the Effect of Tiotropium in Patients With COPD
Brief Title: Dynamic Hyperinflation and Tiotropium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gelb, Arthur F., M.D. (Individual)
Collaborators: Boehringer Ingelheim (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20061693; IIS Boehringer-Ingelheim (Other Grant/Funding Number: Boehringer-Ingelheim and Pfizer); IIS Pfizer (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2017-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tiotropium 18 µg capsule, bronchodilator (Active Comparator): tiotropium 18 µg capsule for 1 month versus placebo. To study bronchodilation and effect following metronome paced hyperventilation and induced dynamic hyperinflation of active tiotropium versus placebo
  Interventions: Drug: Placebo
- 2 (Placebo Comparator): placebo 18ug tiotropium for 1 month
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Procedure/Surgery - tiotropium 18ug capsule daily for 1 month vs placebo to study the effect of trough and peak effect on bronchodilation and effect of metronome paced hyperventilation induced dynamic hyperinflation

SUMMARY:
We will detect dynamic hyperinflation (DH) in 40 COPD (chronic obstructive pulmonary disease) patients with moderately severe disease using metronome paced hyperventilation (MPH) with inspiratory capacity as the primary end point. Hypothesis: Is tiotropium capable of lung volume protecting inspiratory capacity from MPH induced DH vs placebo in a randomized crossover double blinded study.

DETAILED DESCRIPTION:
Study completed with 29 patients studied. Data is being analyzed to evaluate trough and peak effect of 18 µg tiotropium vs placebo on FEV 1 (L)(forced expiratory capacity in one second), inspiratory capacity and functional residual volume. In addition, we will study the effect of 18 µg tiotropium vs placebo on metronome paced hyperventilation induced dynamic hyperinflation. We will also evaluate the effect of tiotropium induced increase in IC (inspiratory capacity) vs extent of emphysema as evaluated on high resolution thin section CT lung

ELIGIBILITY:
Inclusion Criteria:

* Moderately severe COPD patients age 40-85 yr with post 180ug albuterol FEV 1 between 60 and 79% predicted and FEV 1/FVC < 70%.
* Smoking history > 10 pack yr.
* Clinically stable X 6 weeks.
* No oxygen usage.

Exclusion Criteria:

* History of asthma
* Clinically unstable
* Any other significant medical problem precluding full cooperation for study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur F Gelb, MD, Principal Investigator — Arthur F Gelb Medical Corporation; Noe Zamel, MD, Principal Investigator — Mt. Sinai Hosp. Toronto, Univ Toronto Medical Center
Locations (2):
- Arthur F Gelb MD, Lakewood, California, United States
- Noe Zamel MD, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Please see published data

REFERENCES:
- [Background] Gelb AF, Gutierrez CA, Weisman IM, Newsom R, Taylor CF, Zamel N. Simplified detection of dynamic hyperinflation. Chest. 2004 Dec;126(6):1855-60. doi: 10.1378/chest.126.6.1855. PMID 15596684
- [Background] Gelb AF, Taylor CF, McClean PA, Shinar CM, Rodrigues MT, Gutierrez CA, Chapman KR, Zamel N. Tiotropium and simplified detection of dynamic hyperinflation. Chest. 2007 Mar;131(3):690-695. doi: 10.1378/chest.06-1662. PMID 17356081
- [Derived] Gelb AF, Fraser C, Zamel N. Lack of protective effect of tiotropium vs induced dynamic hyperinflation in moderate COPD. Respir Med. 2011 May;105(5):755-60. doi: 10.1016/j.rmed.2010.11.020. Epub 2010 Dec 14. PMID 21159499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with COPD (chronic obstructive pulmonary disease), GOLD (Global Initiative for Chronic Obstructive Lung Disease)Stage 2 were recruited from pulmonary out-patient offices at Mt. Sinai Hosp. Toronto and from Arthur F Gelb MD Lakewood, Calif from June 2009 thru January 2010
Pre-assignment Details: We recruited 30 patients with smoking history >20 pack yr with documented GOLD Stage 2 moderate COPD who were clinically stable for at least 6 weeks prior to the present study and were not on oxygen or oral corticosteroids.
Groups:
- Tiotropium 18 µg Capsule First, Then Placebo; Placebo First, Then Tiotropium Bromide 18 µg: tiotropium 18 µg capsule for 1 month versus placebo. To study bronchodilation and effect following metronome paced hyperventilation and induced dynamic hyperinflation of active tiotropium versus placebo
Period: Period: First Intervention
Arm/Group | Tiotropium 18 µg Capsule First, Then Placebo | Placebo First, Then Tiotropium Bromide 18 µg
Started | 15 (randomized cross over study) | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Period: Second Intervention
Arm/Group | Tiotropium 18 µg Capsule First, Then Placebo | Placebo First, Then Tiotropium Bromide 18 µg
Started | 15 | 14
29 Days | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive placebo first and Tiotropium first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 23
  Canada | 6
Average participant age +/- SD [Mean (Standard Deviation); unit: years] — One patient was dropped due to a protocol violation.
  years | 70 (9)
FVC (forced vital capacity) [Mean (Standard Deviation); unit: liters] — forced vital capacity (observed)
  liters
    FVC (L) | 2.9 (1.2)
    FVC (L) post 180 µg albuterol sulfate MDI | 3.3 (1.2)
FVC [Mean (Standard Deviation); unit: percentage of liters expected] — Forced vital capacity - % predicted
  percentage of liters expected
    FVC percent of liters predicted | 86 (17)
    FVC post 180 µg albuterol percent of ltrs predict | 95 (16)
FEV1(L) (forces expiratory volume) observed [Mean (Standard Deviation); unit: liters] — Forced expiratory volume in 1s, observed
  liters
    FEV1(L) | 1.6 (0.6)
    FEV1(L) post 180 ug albuterol sulfate MDI | 1.8 (0.6)
FEV1 (L) percent predicted [Mean (Standard Deviation); unit: percentage of liters expected] — forced vital capacity (L) - percent predicted
  percentage of liters expected
    FEV1 percent liters predicted | 61 (69)
    FEV1 percent liters predicted post albuterol | 8 (6)
FEV1/FVC percentage [Mean (Standard Deviation); unit: percentage of liters expected] — forced expiratory volume in 1s/forced vital capacity - percent
  percentage of liters expected | 56 (8)
SGaw (Lps/cmH2O/L) (specific airway conductance) [Mean (Standard Deviation); unit: Lps/cmH2O/L] — specific airway conductance (observed)
  Lps/cmH2O/L | 0.10 (0.08)
FRC (L) (functional residual capacity) observed [Mean (Standard Deviation); unit: liters] — functional residual capacity - observed
  liters | 3.9 (0.8)
FRC percent of liters predicted [Mean (Standard Deviation); unit: percentage of liters predicted] — functional residual capacity percent of liters predicted
  percentage of liters predicted | 138 (29)
RV (L) (residual volume) observed [Mean (Standard Deviation); unit: liters] — residual volume (liters) observed
  liters | 2.9 (0.1)
RV (L) - % predicted [Mean (Standard Deviation); unit: percentage] — residual volume (L) - percent predicted
  percentage | 131 (37)
TLC (L) (total lung capacity) observed [Mean (Standard Deviation); unit: liters] — total lung capacity - observed
  liters | 5.9 (1.3)
TLC Percent of liters predicted [Mean (Standard Deviation); unit: percentage of liters predicted] — total lung capacity - percent of liters predicted
  percentage of liters predicted | 109 (16)
D(L)CO(SB) - ml/min/mmHg observed (Single-breath diffusing capacity ) [Mean (Standard Deviation); unit: ml/min/mmHg] — Single-breath diffusing capacity (ml/min/mmHg)observed
  ml/min/mmHg | 14 (5)
D(L)CO(SB) - ml/min/mmHg % predicted [Mean (Standard Deviation); unit: ml/min/mmHg] — single-breath diffusing capacity - ml/min/mmHg - percent predicted
  ml/min/mmHg | 69 (23)

OUTCOME MEASURES:

1. Primary Outcome: Bronchodilator Response:Peak FEV1(L)(Forced Expiratory Volume in One Second)-
Description: Lung function studies (mean +/- SD): peak FEV1 (+2h) after 30 days of placebo or tiotropium in 29 moderate COPD patients. FEV1 = Forced expiratory volume in one second
Time Frame: 30 days
Population: Lung function studies (mean +/- SD): peak FEV1 (+2h) after 30 days of placebo or tiotropium in 29 moderate COPD patients. FEV1 = Forced expiratory volume in one second
Measure: Mean (Standard Deviation); unit: liters
Groups:
- Placebo; Tiotropium: Includes groups randomized to receive placebo first and Tiotropium first.
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 29 | 29
liters | 1.74 (0.58) | 1.82 (0.59)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Mean difference of Peak FEV1 of tiotropium minus placebo. 29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis — a priori threshold for statistical significance: p<0.05

2. Secondary Outcome: Extent of Lung CT Scored Emphysema and and Lung Function of FEV1(l) After Tiotropium
Description: Correlation between improved lung function after tiotropium and extent of lung CT scored emphysema with respect to FEV 1; correlation of tiotropium induced bronchodilation and extent of lung ct scored emphysema; measures include increase in FEV1 from baseline to peak tiotropium
Time Frame: baseline to 30 days
Population: High-resolution, thin-section scans of the lung were obtained from a subset of 19 patients.
Measure: Mean (Standard Deviation); unit: percentage of lung tissue
Groups:
- Lung CT Scored Emphysema and FEV1: Extent of lung CT scored emphysema and and lung function of FEV1(l) after tiotropium
Arm/Group | Lung CT Scored Emphysema and FEV1
Number analyzed (Participants) | 19
percentage of lung tissue | 13.68 (18.84)
Statistical Analysis 1: Comparison: Lung CT Scored Emphysema and FEV1; Correlation between improved lung function after tiotropium and extent of lung CT scored emphysema with respect to ratio functional residual capacity divided by total lung capacity. Specifically, correlation of tiotropium induced bronchodilation and extent of lung ct scored emphysema; measure includes change in FEV1 post tiotropium; Test type: Superiority or Other; p = 0.96, Spearman rho — A priori threshold for statistical significance: p=0.05; Spearman rho = 0.19

3. Primary Outcome: Bronchodilator Response:Peak FRC (L) (Functional Residual Capacity)
Description: Lung function studies (mean +/- SD): peak FRC after 30 days (+2h) of placebo or tiotropium in 29 moderate COPD patients.
Time Frame: 30 days
Population: Includes groups randomized to receive placebo first and Tiotropium first.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 29 | 29
Liters | 3.80 (0.79) | 3.72 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Mean difference of Peak FRC in tiotropium minus placebo. 29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = 0.318, Mixed Models Analysis — A priori threshold for statistical significance: p<0.05

4. Primary Outcome: Bronchodilator Response: Peak FVC (L) (Forced Vital Capacity)- Tiotropium and Placebo
Description: Lung function studies (mean +/- SD) of peak forced vital capaciy (L) after 30 days (+2h) of tiotropium versus placebo in 29 moderate COPD patients. Forced vital capacity - liters
Time Frame: 30 days
Population: Peak FVC after 30 days (+2h) of tiotropium versus placebo in 29 moderate COPD patients.
Measure: Mean (Standard Deviation); unit: liters
Groups:
- Tiotropium 18 µg Capsule, Bronchodilator: Includes groups randomized to receive placebo first and Tiotropium first.
Arm/Group | Placebo | Tiotropium 18 µg Capsule, Bronchodilator
Number analyzed (Participants) | 29 | 29
liters | 3.17 (1.13) | 3.27 (1.16)
Statistical Analysis 1: Comparison: Placebo; Mean difference of Peak FVC of tiotropium minus placebo.29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = 0.078, Mixed Models Analysis — Statistical significance was p < 0.05

5. Secondary Outcome: IC (Inspiratory Capacity, L) Post Mph (Metronome Paced Hyperventilation) Induced dh (Dynamic Hyperinflation) After Tiotropium and Extent of Lung CT Scored Emphysema
Description: Correlation between change in inspiratory capacity (L) post metronome paced hyperventilation induced dynamic hyperinflation and extent of lung ct scored emphysema
Time Frame: baseline to 30 days
Population: Analysis was carried out per protocol
Measure: Mean (Standard Deviation); unit: percentage of lung tissue
Groups:
- Lung CT Scored Emphysema and IC: Extent of lung CT scored emphysema (percent of lung) and lung function of IC (inspiratory capacity, L) after tiotropium.
Arm/Group | Lung CT Scored Emphysema and IC
Number analyzed (Participants) | 19
percentage of lung tissue | 13.68 (18.84)
Statistical Analysis 1: Comparison: Lung CT Scored Emphysema and IC; Correlation between improved lung function after tiotropium and extent of lung CT scored emphysema with respect to ratio functional residual capacity divided by total lung capacity. Specifically, correlation of tiotropium induced bronchodilation and extent of lung ct scored emphysema (19 patients); measures include change in IC at trough tiotropium; Test type: Superiority or Other; p = 0.4, Spearman rho; Spearman rho = -0.26

6. Primary Outcome: Bronchodilator Response: Peak IC (L) - (Inspiratory Capacity) - Tiotropium Versus Placebo
Description: Lung function studies (mean +/- SD) - Peak inspiratory capacity after 30 days (+2h)of tiotropium versus placebo in 29 moderate COPD patients. Inspiratory capacity- liters
Time Frame: 30 days
Population: Net change in lung function studies (mean +/- SE) from baseline to trough (-1h) and peak (+2h) after 30 days of tiotropium versus placebo in 29 moderate COPD patients.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 29 | 29
liters | 2.12 (0.82) | 2.24 (0.80)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Mean difference of Peak IC of tiotropium minus placebo.29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = 0.067, Mixed Models Analysis — A priori threshold for statistical significance: p<0.05

7. Primary Outcome: Bronchodilator Response: Peak FRC/TLC Percentage (Functional Residual Capacity(L)/Total Lung Capacity(L) - Tiotropium or Placebo
Description: Lung function studies (mean +/- SD) peak Peak FRC/TLC after 30 days (+2h)of tiotropium versus placebo in 29 moderate COPD patients. Functional residual capacity/total lung capacity - percentage
Time Frame: 30 days
Population: Lung function studies (mean +/- SD) peak Peak FRC/TLC after 30 days (+2h)of tiotropium versus placebo in 29 moderate COPD patients. Functional residual capacity/total lung capacity - percentage
Measure: Mean (Standard Deviation); unit: percentage of FRC/TLC
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 29 | 29
percentage of FRC/TLC | 0.65 (0.10) | 0.66 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Mean difference of Peak FRC/TLC of tiotropium minus placebo. 29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = 0.615, Regression, Logistic — A priori threshold for statistical significance: p<0.05

8. Primary Outcome: Bronchodilator Response: Peak TLC (L) (Total Lung Capacity)- Tiotropium or Placebo
Description: Net change in lung function studies (mean +/- SE) from baseline to trough (-1h) and peak (+2h) after 30 days of tiotropium versus placebo in 29 moderate COPD patients. Total lung capacity - liters
Time Frame: 30 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 29 | 29
liters | 5.91 (1.22) | 5.82 (1.35)
Statistical Analysis 1: Comparison: Placebo; 29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = 0.325, Mixed Models Analysis — Statistical significance was p<0.05

9. Primary Outcome: Bronchodilator Response: Trough FEV1 (L)- (Forced Expiratory Volume) Tiotropium Versus Placebo
Description: Lung function studies Trough FEV1(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients. Forced expiratory volume in 1s (liters)
Time Frame: 30 days
Population: Lung function studies Trough FEV1(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 29 | 29
liters | 1.68 (0.54) | 1.71 (0.56)
Statistical Analysis 1: Comparison: Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.345, Mixed Models Analysis

10. Primary Outcome: Bronchodilator Response: Trough FRC (L)- Tiotropium Versus Placebo
Description: Lung function studies Trough FRC(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients. Functional residual capacity(liters)
Time Frame: 30 days
Population: Lung function studies Trough FRC(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients. Functional residual capacity(liters)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 29 | 29
liters | 3.84 (0.84) | 3.66 (0.88)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Mean difference of Trough FRC(L) in tiotropium minus placebo. 29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = 0.068, Mixed Models Analysis — A priori threshold for statistical significance: p<0.05

11. Primary Outcome: Bronchodilator Response: Trough FVC (L)- (Forced Vital Capacity) Tiotropium Versus Placebo
Description: Lung function studies Trough FVC(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients
Time Frame: 30 days
Population: Lung function studies Trough FVC(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 29 | 29
liters | 3.12 (1.10) | 3.15 (1.13)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Mean difference of trough FVC in tiotropium minus placebo. 29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = 0.589, Mixed Models Analysis — A priori threshold for statistical significance: p<0.05

12. Primary Outcome: Bronchodilator Response: Trough IC (L) Inspiratory Capacity - Tiotropium Versus Placebo
Description: Lung function studies (Trough IC(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients Trough inspiratory capacity- liters
Time Frame: 30 days
Population: Lung function studies (Trough IC(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients Trough inspiratory capacity- liters
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 29 | 29
liters | 2.17 (0.77) | 2.11 (0.83)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Mean difference of Trough IC of tiotropium minus placebo. 29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = 0.922, Mixed Models Analysis — A priori threshold for statistical significance: p<0.05

13. Primary Outcome: Bronchodilator Response: Trough FRC/TLC (Functional Residual Capacity/Total Lung Capacity)- Tiotropium Versus Placebo
Description: Lung function studies Trough FRC/TLC(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients Trough Functional residual capacity/total lung capacity - percentage
Time Frame: 30 days
Population: Lung function studies Trough FRC/TLC(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients Trough Functional residual capacity/total lung capacity - percentage
Measure: Mean (Standard Deviation); unit: percentage of FRC/TLC
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 29 | 29
percentage of FRC/TLC | 0.64 (0.09) | 0.62 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Mean difference of Trough FRC/TLC of tiotropium minus placebo. 29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = -0.02, Mixed Models Analysis — A priori threshold for statistical significance: p<0.05

14. Primary Outcome: Bronchodilator Response: Trough TLC (L) (Total Lung Capacity)- Tiotropium Versus Placebo
Description: Lung function studies Trough TLC(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients
Time Frame: 30 days
Population: Lung function studies Trough TLC(mean +/- SD) after 30 days(-1h) of tiotropium versus placebo in 29 moderate COPD patients
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Tiotropium
Number analyzed (Participants) | 29 | 29
liters | 5.99 (1.18) | 5.86 (1.25)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium; Mean difference of Trough TLC (L) of tiotropium minus placebo. 29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = -0.13, Mixed Models Analysis — A priori threshold for statistical significance: p<0.05

15. Primary Outcome: IC (Inspiratory Capacity L)and Metronome Paced Hyperventilation-induced Dynamic Hyperinflation in Tiotropium Cohort Versus Placebo and Baseline
Description: IC measurement before and after metronome paced hyperventilation-induced dynamic hyperinflation at baseline and in tiotropium and placebo groups. Measure ratio of functional residual capacity divided by total lung capacity at baseline and after 30 days of tiotropium versus placebo
Time Frame: baseline and 30 days (+2h) post dose
Population: Inspiratory capacity (IC) (mean +/- SD) from baseline and after 30 days of tiotropium versus placebo in 29 moderate COPD patients.
Measure: Mean (Standard Deviation); unit: liters
Groups:
- Before DH (Dynamic Hyperinflation): IC (inspiratory capacity) before and after metronome paced hyperventilation and induced dynamic hyperinflation at baseline;
- After DH (Dynamic Hyperinflation: IC (inspiratory capacity) before and after metronome paced hyperventilation induced dynamic hyperinflation post 30 days plus 2h placebo
Arm/Group | Before DH (Dynamic Hyperinflation) | After DH (Dynamic Hyperinflation
Number analyzed (Participants) | 29 | 29
liters
  Baseline IC (inspiratory capacity) | 2.09 (0.83) | 1.76 (0.70)
  Placebo IC | 2.17 (0.82) | 1.80 (0.70)
  Tiotropium IC | 2.24 (0.80) | 1.80 (0.74)
Statistical Analysis 1: Comparison: Before DH (Dynamic Hyperinflation) vs After DH (Dynamic Hyperinflation; Change in IC before and after dynamic hyperinflation. 29 patients needed to achieve a power of 80% at a significant alpha level of 5% using projected sample inspiratory capacity of 2.23+/- 0.5L post tiotropium compared to baseline inspiratory capacity 2.0+/-0.5L; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — A priori threshold for statistical significance: p<0.05

16. Primary Outcome: TLC (L) Before and After Metronome Paced Hyperventilation Induced Dynamic Hyperinflation in Tiotropium Cohort Versus Placebo
Description: Total lung capacity before and after metronome paced hyperventilation induced dynamic hyperinflation in tiotropium cohort versus placebo. Difference between TLC measured at one hour before intervention & 2 hrs. after after 30 days of treatment with either placebo or tiotropium
Time Frame: one hour before intervention & 2 hrs. after after 30 days
Population: lung function studies (mean +/- SE) from baseline to trough (-1h) and peak (+2h) after 30 days of tiotropium versus placebo in 29 moderate COPD patients.
Measure: Mean (Standard Deviation); unit: liters
Groups:
- 2h Post Placebo TLC(L): total lung capacity (L) following metronome paced hyperventilation induced dynamic hyperinflation post 30 days plus 2h placebo
- TLC (L) 2h Post Tiotropium: Total Lung Capacity (L)following metronome paced hyperventilation induced dynamic hyperinflation post 30 days plus 2h tiotropium
Arm/Group | 2h Post Placebo TLC(L) | TLC (L) 2h Post Tiotropium
Number analyzed (Participants) | 29 | 29
liters
  Before DH (dynamic hyperinflation) | 5.96 (1.22) | 5.84 (1.35)
  After DH | 5.84 (1.13) | 5.78 (1.14)
Statistical Analysis 1: Comparison: 2h Post Placebo TLC(L) vs TLC (L) 2h Post Tiotropium; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis — Total lung capacity was similar in all groups and was not significant

17. Secondary Outcome: Extent of Lung CT Scored Emphysema and and Lung Function of FRC/TLC (Functional Residual Capacity(L)/Total Lung Capacity (L) After Tiotropium
Description: Correlation between improved lung function after tiotropium and extent of lung CT scored emphysema with respect to ratio functional residual capacity divided by total lung capacity. Specifically, correlation of tiotropium induced bronchodilation and extent of lung ct scored emphysema
Time Frame: baseline to trough tiotropium
Population: High resolution, thin-section scans of the lung were obtained in a subset of 19 patients.
Measure: Mean (Standard Deviation); unit: percentage of lung tissue
Groups:
- Lung CT Scored Emphysema and FRC/TLC: Extent of lung CT scored emphysema (percent of lung) and lung function of FRC/TLC (functional residual capacity(L)/total lung capacity (L) after tiotropium
Arm/Group | Lung CT Scored Emphysema and FRC/TLC
Number analyzed (Participants) | 19
percentage of lung tissue | 13.68 (18.84)
Statistical Analysis 1: Comparison: Lung CT Scored Emphysema and FRC/TLC; Correlation between improved lung function after tiotropium and extent of lung CT scored emphysema with respect to ratio functional residual capacity divided by total lung capacity. Specifically, correlation of tiotropium induced bronchodilation and extent of lung ct scored emphysema; Test type: Superiority or Other; p = 0.36, Spearman rho — A priori threshold for statistical significance: p= 0.05; Spearman rho = -0.26

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Tiotropium Bromide 18 µg, Capsule,: tiotropium 18 µg capsule for 1 month. To study bronchodilation and effect following metronome paced hyperventilation and induced dynamic hyperinflation of active tiotropium. (30 enrolled subjects, one drop-out)
- Placebo: Adverse events after placebo. (30 enrolled subjects, one drop-out)
Arm/Group | Tiotropium Bromide 18 µg, Capsule, | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No